CLINICAL TRIAL: NCT04976140
Title: A Prospective, Open, Dose-escalation, Multi-center, Phase 1/2a Trial to Evaluate the Safety, Tolerability and to Explore the Efficacy of PN-101 in Patients With Refractory Polymyositis or Dermatomyositis
Brief Title: Allogeneic Mitochondria (PN-101) Transplantation for Refractory Polymyositis or Dermatomyositis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paean Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PN-101-101
Record Dates: First submitted 2021-07-01; First posted 2021-07-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: mitochondria
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): The investigational product is intravenously administered according to the planned dose.
  Interventions: Biological: PN-101
- Intermediate dose group (Experimental): The investigational product is intravenously administered according to the planned dose.
  Interventions: Biological: PN-101
- High dose group (Experimental): The investigational product is intravenously administered according to the planned dose.
  Interventions: Biological: PN-101

INTERVENTIONS:
Biological: PN-101 — PN-101: Mitochondria isolated from Allogeneic Umbilical Cord-derived Mesenchymal Stem Cells.
  3 or 6 subjects are enrolled in each dose group in line with the traditional 3+3 rule-based method, and the investigator intravenously administers a single-dose of the investigational product according to the planned dose.

SUMMARY:
To determine the maximum tolerated dose (MTD) based on the safety and tolerability after single-dose administration of PN-101 in patients with refractory polymyositis or dermatomyositis. To explore the efficacy after single-dose administration of PN-101 in patients with refractory polymyositis or dermatomyositis.

DETAILED DESCRIPTION:
This Phase 1/2a clinical trial involves patients diagnosed with refractory polymyositis or dermatomyositis.

The initial safety assessment is conducted, including development of DLT in subjects up to Week 2 after the investigational product administration.

[DLT assessment criteria and method]

* Low dose or intermediate dose level

  1. No DLT developing in the initially enrolled 3 subjects (0/3): Increase the dose to the next dose group
  2. DLT developing 1 of 3 subjects (1/3): Enroll 3 additional subjects at the same dose group and then assess DLT, and ① DLT developing in 1 out of total 6 subjects (1/3+0/3; 1/6): Increase the dose to the next dose group ② DLT developing in ≥ 2 out of total 6 subjects (≥ 2/6): In case of the low dose level, the trial is discontinued without MTD determination. In case of the intermediate dose level, MTD is assessed at the low dose which is a one lower dose level
* High dose level

  1. No DLT developing in the initially enrolled 3 subjects (0/3): Declare as the MTD
  2. DLT developing 1 of 3 subjects (1/3): Enroll 3 additional subjects at the same dose group and then assess DLT, and ① DLT developing in 1 out of total 6 subjects (1/3+0/3; 1/6): Declare as the MTD ② DLT developing in ≥ 2 out of total 6 subjects (≥ 2/6): Assess MTD at the intermediate dose which is the one lower dose level

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 years or more
2. A subject who is diagnosed with polymyositis or dermatomyositis and satisfies all of the followings

   * Clinical profile: Slowly progressing clinical profile with symmetrical and apparent muscular weakness confirmed at the proximal muscle (in case of dermatomyositis, clinical findings related with characteristic skin symptoms*)

     * Gottron's papules or sign, erythema purpura, poikiloderma, calcinosis cutis, etc.
   * Serum test: Serum creatine kinase (CK) elevated (CK ≥ 1.3 × upper limit of normal (ULN)) or serum myositis-specific antibodies (MSA) positive
   * Electromyography (EMG): Presence of a finding that indicates myopathy
3. Baseline (prior to the investigational product administration) manual muscle testing-8 (MMT-8) result < 125/150 (bilaterally), and at least 2 of the following International Myositis and Clinical Studies Group (IMACS) core set results

   * Physician global disease activity [visual analogue scale (VAS)] ≥ 2 cm
   * Patient global disease activity [VAS] ≥ 2 cm
   * Health assessment questionnaire (HAQ) disability assessment ≥ 0.25
   * 1 or more items with the serum muscle enzyme > 1.3 × ULN
   * Global extramuscular disease activity [VAS] > 1 cm
4. A subject with the drug treatment history of polymyositis or dermatomyositis for ≥ 8 weeks, who cannot receive the conventional treatment due to being refractory or for a side effect and adverse event, and has received glucocorticosteroids at an intermediate dose (prednisone 0.5 mg/kg/day or equivalent) or higher for at least 4 weeks alone or in combination
5. A subject who fully understands the trial and provided voluntary written consent to take part in the trial

Exclusion Criteria:

1. A subject with clear muscular damage, with the VAS-based myositis damage index (MDI) of ≥ 5 at screening
2. A subject with the following medical history or surgical history

   * A surgical operation history within 12 weeks of screening
   * Malignant tumor within 5 years of screening (excluding a subject who passed 3 years or more from complete recovery of cervical cancer or skin squamous cell carcinoma)
3. A patient with severe respiratory muscular weakening or interstitial pulmonary disease (a patient who has no moderate or severe dyspnea and has stable interstitial pneumonia may participate)
4. A patient with the following comorbidity at screening

   * Acute viral infection or severe infection
   * Active hepatitis B (e.g.: HBsAg positive and HBV DNA detected) or hepatitis C (e.g.: Anti-HCV positive and HCV RNA [qualitatively] detective)
   * Human Immunodeficiency virus (HIV) positive
   * Findings of muscular inflammation or myopathy other than the indication (inclusion body myositis (IBM), drug-induced myopathy, amyloid myopathy, myotonic dystrophy, etc.)
   * Autoimmune disease such as rheumatoid arthritis (RA), systemic lupus erythematosus, psoriatic arthritis, etc. (however, in case of the overlap syndrome, a subject may participate if diseases other than inflammatory myositis are stable and myositis is thought to be due to inflammatory myositis.)
   * Findings of cardiac disorder such as moderate or severe heart failure (New York Heart Association Class III/IV) or QT corrected interval prolonged
   * Serious disease that may affect this study, at the discretion of the investigator (neurological disorder, cardiovascular disorder, uncontrolled blood pressure or diabetes, etc.)
5. Hematological, renal and hepatic dysfunction based on the following laboratory findings at screening

   * Glomerular filtration rate (GFR)* < 45 mL/min

     *eGFR (mL/min/1.73m^2) = 175 × (serum creatinine concentration (mg/dL))^-1.154 × (age)^-0.203 × (0.742 in female) [modification of diet in renal disease (MDRD) formula]
   * Hemoglobin < 10 g/dL
   * White blood cell (WBC) count < 3.0×10^9/L
   * Absolute neutrophil count (ANC) < 1.5×10^9/L (1500/mm^3)
   * Platelet count < 100×10^9/L
   * AST and ALT > 2.5 × ULN (except for the elevation due to muscle enzyme at the discretion of the investigator)
   * Alkaline phosphatase (ALP) > 2.5 × ULN
   * Total bilirubin > 1.5 × ULN (> 3 × ULN, in case of Gilbert's syndrome)
   * Thyroid stimulating hormone level exceeding the normal range (however, if the level exceeds the normal range due to the study indication at the discretion of the investigator, the subjects are allowed to enroll.)
6. A subject with a difficulty in the efficacy assessment including the muscular strength assessment during the trial
7. A subject who is determined to require prohibited concomitant treatment during the trial
8. Pregnant woman and lactating mother or woman of childbearing potential and man who is planning to have a child or not willing to practice acceptable contraception* during the trial

   *Hormonal contraception, intrauterine device or intrauterine system implant, double barrier method (use of both male condom and occlusive cap (contraceptive diaphragm or cervical cap) along with spermicide), surgical sterilization procedure/operation (vasectomy, tubal ligation, etc.)
9. Participation in other clinical trial and administration of an investigational product or application of an investigational device within 4 weeks or half-life x 5 (whichever is longer) prior to screening
10. A subject who is otherwise ineligible for this trial, at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity(DLT) | 2 weeks after IP administration
  Assessment of DLT for each dose group up to 2 weeks after the IP administration.
  Severity will be graded according to CTCAE, Version 5.0.
International Myositis And Clinical Studies group-Total Improvement Score(IMACS-TIS) | 12 weeks after the IP administration
  Assessment of IMACS-TIS at Week 12 after the IP administration. Total Improvement Score (TIS) based on absolute percentage change is assessed scale 0 to 100. Higher score indicates greater improvement.

SECONDARY OUTCOMES:
International Myositis And Clinical Studies group-Total Improvement Score(IMACS-TIS) | 4 weeks after the IP administration
  Assessment of IMACS-TIS at week 4 after the IP administration. Total Improvement Score (TIS) based on absolute percentage change is assessed scale 0 to 100. Higher score indicates greater improvement.
International Myositis And Clinical Studies group-Total Improvement Score(IMACS-TIS) | 8 weeks after the IP administration
  Assessment of IMACS-TIS at week 8 after the IP administration. Total Improvement Score (TIS) based on absolute percentage change is assessed scale 0 to 100. Higher score indicates greater improvement.
Response rate of IMACS-TIS | 12 weeks after the IP administration
  Proportion of subjects with the IMACS-TIS ≥ 20 at week 12 after the IP administration.
Changes of Core Set Activity Measures(CSAM) | Visit 2(Day 1), Visit 5(4 weeks), Visit 6(8 weeks), Visit 7(12 weeks)
  Changes in CSAM for the IMACS assessed at week 4, week 8 and week 12 after the IP administration from the baseline (Visit 2).
Changes of Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) | Visit 2(Day 1), Visit 5(4 weeks), Visit 6(8 weeks), Visit 7(12 weeks)
  Changes in CDASI assessed at week 4, week 8 and week 12 after the IP administration from the baseline (Visit 2) for dermatomyositis only.
Changes of Peak Pruritus Numeral Rating Scale(PPNRS) | Visit 2(Day 1), Visit 5(4 weeks), Visit 6(8 weeks), Visit 7(12 weeks)
  Changes in PPNRS assessed at week 4, week 8 and week 12 after the IP administration from the baseline (Visit 2) for dermatomyositis only. The intensity of pruritis is assessed on a patient reported scale 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Eunyoung Lee, MD, Principal Investigator — Seoul National University College of Medicine; Daehyun Yoo, MD, Principal Investigator — Hanyang University College of Medicine; Hyunsook Kim, MD, Principal Investigator — Soonchunhyang University College of Medicine
Locations (3):
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No